CLINICAL TRIAL: NCT01337648
Title: Radiation Biodosimetry in Children Undergoing Total Body Irradiation
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, John Baker, Professor of Surgery/Cardiothoracic/Research, Medical College of Wisconsin
Other Study IDs: RadBio-10/191
Record Dates: First submitted 2011-03-02; First posted 2011-04-19 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Total-body Irradiation; Hematopoietic Stem Cell Transplant
Keywords: Fecal biomarkers; Radiation biodosimetry; Total-body irradiation (TBI); Hematopoietic stem cell transplantation; Gene expression profiles; Fecal metabolites

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TBI prior to stem cell transplantation

SUMMARY:
The purpose of this study is to develop fecal tests that will determine the extent of radiation exposure in patients undergoing radiation treatment for cancer. This project will determine whether fecal biomarkers can be used to diagnose exposure to radiation.

DETAILED DESCRIPTION:
Patients undergoing TBI as part of a hematopoietic stem cell transplant (HSCT) will have feces collected for use in the validation and refinement of new methods for rapid radiation biodosimetry. The stool samples will be collected before, and at defined times after TBI. Stool sampling will occur in the same manner that it does during routine patient care during HSCT.

ELIGIBILITY:
Inclusion Criteria:

* All races are eligible
* 2 years to 21 years old
* Must be undergoing hematopoietic stem cell transplantation (either autologous or allogeneic) in conjunction with a conditioning regimen that includes total-body irradiation (TBI) (single or multiple fraction).

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients undergoing Total Body Irradiation (TBI) preceding hematopoietic stem cell transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2010-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
To describe changes in gene expression associated with exposure to radiation | prior to TBI treatment (baseline) and up to 2 weeks following the last dose of TBI
  Changes in gene expression will be measured as abundance of RNA levels relative to the weight of feces

CONTACTS AND LOCATIONS:
Overall Officials: John Baker, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States